CLINICAL TRIAL: NCT02796898
Title: A Phase 1b/2, Open-Label, Dose Escalation Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of SM88 in Patients With Prostate Cancer
Brief Title: Study of the Efficacy, Safety, and Pharmacokinetics of SM88 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tyme, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tyme 2016b
Record Dates: First submitted 2016-05-30; First posted 2016-06-13 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Prostate Cancer; Rising Prostate Specific Antigen (PSA)
Keywords: Prostate Cancer; PSA; Androgen Deprivation Therapy (ADT)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — racemetyrosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treated Group (Experimental): SM88 is a combination therapy consisting of 4 agents. One agent, the tyrosine isomer will be increased in each of 2 dose cohorts as follows:
  Cohort 1:
  * Tyrosine isomers - 230 mg qd
  * Phenytoin - 50 mg qd.
  * Methoxsalen - 10 mg qd
  * Sirolimus - 0.5 mg qd
  Cohort 2:
  Cohort 2 has increasing tyrosine isomer from q.d. to b.i.d.
  Expansion Cohort:
  The optimum dose will be expanded in 2nd stage of the study to 30 subjects.
  Interventions: Drug: SM88 (Cohort 1); Drug: SM88 (Cohort 2)

INTERVENTIONS:
Drug: SM88 (Cohort 1) — * Tyrosine Isomers - 230 mg qd
  * Phenytoin - 50 mg qd.
  * Methoxsalen - 10 mg qd
  * Sirolimus - 0.5 mg qd
  Other Names: SM88
Drug: SM88 (Cohort 2) — * Tyrosine Isomers - 460 mg (230 mg bid)
  * Phenytoin - 50 mg qd
  * Methoxsalen - 10 mg qd
  * Sirolimus - 0.5 mg qd
  Other Names: SM88

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics, and efficacy of SM88 in patients with prostate cancer

DETAILED DESCRIPTION:
This is an open-label, multi-center, dose-escalating, dose-expansion study of SM88 in patients with prostate cancer. This study includes 2 phases, a dose-escalation phase that includes PK evaluation, and a dose-expansion phase.

During the first stage, at up to 2 institutions, up to 2 cohorts of 1 to 6 patients each will be enrolled.

During the second stage, the dose selected for evaluation from the Phase 1b will be administered for a total of 30 evaluable patients (inclusive of those treated at the same dose during the dose selection phase) for 6 cycles or until unacceptable toxicity, disease progression, or until any of the treatment discontinuation criteria are met.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥18 years of age.
2. Histologically or cytologically confirmed prostate cancer (patients with neuroendocrine carcinoma of the prostate are excluded).
3. Documented PSA progression. Pre-enrollment PSA progression will be as defined by the PCWG3 criteria, e.g. 3 values, increasing, each >7 days apart.
4. ECOG performance status ≤1
5. Life expectancy >3 months, in the judgment of the investigator.
6. Adequate organ function defined as follows:

   1. Hematologic: Platelets ≥100 x 109 /L; Absolute Neutrophil Count (ANC) ≥1.5 x 109/L (without platelet transfusion or growth factors within the 7 days prior to the screening laboratory assessment)
   2. Hepatic: aspartate transaminase (AST)/alanine transaminase (ALT) ≤2.5 x upper limit of normal (ULN); total or conjugated bilirubin ≤1.5 x ULN
   3. Renal: serum creatinine ≤1.5 x ULN or creatinine clearance (CrCl) ≥60 mL/min as calculated by the Cockroft-Gault method
7. Coagulation: International normalized ratio (INR) ≤1.2
8. With or without one prior line of chemotherapy
9. With or without prior or current ADT or hormone based therapy (up to 2 lines total)
10. Cannot tolerate standard chemotherapy, hormone based therapy or ADT, or elects to opt out of standard therapies.
11. Patients who are on ADT prior to the study need not discontinue such therapy during the study, but the use of ADT during the study must be documented.
12. All acute toxic effects of any prior antitumor therapy resolved to Grade ≤1 before baseline, with the exception of alopecia (Grade 1 or 2 permitted) and neurotoxicity (Grade 1 or 2 permitted)
13. Male patients of fertile potential who engage in heterosexual intercourse with female partners of childbearing potential must agree to use highly effective contraception while enrolled in the study and for at least 6 months following the last dose of study drug. Highly effective birth control methods include the following (the patient should choose 2 to be used with their partner):

    1. Oral, injectable, or implanted hormonal contraceptives
    2. Condom with a spermicidal foam, gel, film, cream, or suppository
    3. Occlusive cap (diaphragm or cervical/vault cap) with a spermicidal foam, gel, film, cream, or suppository
    4. Intrauterine device
    5. Intrauterine system (for example, progestin-releasing coil)
    6. Vasectomized male (as determined by the investigator)
14. Able and willing to provide written informed consent to participate in this study

Exclusion Criteria:

1. PSA minimum starting value <1 ng/mL at trial entry.
2. Metastatic disease as detected on bone scan, Computed Tomography (CT), Magnetic Resonance Imaging (MRI), or CT-positron emission tomography (PET) beyond the prostate or post-surgical prostate area.
3. Any screening laboratory, electrocardiogram (ECG), or other findings that, in the opinion of the investigator or the sponsor, indicate an unacceptable risk for the patient's participation in the study.
4. History or evidence of any clinically significant disorder, condition, or disease that, in the opinion of the investigator or medical monitor would pose a risk to the patient's safety or interfere with the study evaluations, procedures, or completion. Examples include intercurrent illness such as active uncontrolled infection, active or chronic bleeding event within 28 days of baseline, uncontrolled cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.
5. History of a concurrent or second malignancy, except for adequately treated local basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, adequately treated Stage 1 or 2 cancer currently in complete remission; or any other cancer that has been in complete remission for ≥5 years
6. Local therapy such as radiation or surgery within 8 weeks of study baseline.
7. Current use of a prohibited medication (see Section 8.5) or requires any of these medications during treatment phase
8. Major surgery, defined as any surgical procedure that involves general anesthesia and a significant incision (i.e., larger than that required for placement of central venous access, percutaneous feeding tube, or biopsy) within 28 days of the first dose of study drug
9. Minor surgical procedures within 7 days of baseline, or not yet recovered from prior surgery
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of any of the components of SM88, e.g. cirrhosis
11. Known human immunodeficiency (HIV) virus infection
12. Hepatitis B surface antigen (HBsAg) positive
13. Hepatitis C virus (HCV) antibody positive
14. Have previously been enrolled in this study or any other study investigating SM88
15. History of any drug allergies or significant adverse reactions to any of the components of SM88.
16. Are currently enrolled in, or have discontinued within 30 days of screening, from a clinical trial involving an investigational product or non-approved use of a drug or device.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06; Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
The dose limiting toxicity (DLT), and maximum tolerated dose (MTD) or minimum effective optimum dose of SM88, when 2 dose levels of SM88 are evaluated. | Six months
  During 4 days of single dose PK evaluations [Phase 1b only], and six 4-week treatment cycles, we will determine if patients in consecutive cohorts experience any dose limiting toxicity to determine MTD, or a complete response with no DLTs observed to determine the optimum dose.

SECONDARY OUTCOMES:
Single dose pharmacokinetics (PK) of tyrosine based isomer alone and as a component of SM88 in patients with prostate cancer. | Six months
  After a single dose of tyrosine based isomer alone on PK Day 1, and a single dose of SM88 on PK Day 3, the plasma concentrations of tyrosine isomers in patients with prostate cancer will be assayed.
Multi-dose PK of the individual isomers of tyrosine. | Six months
  The plasma concentrations of tyrosine isomers associated with morning and evening doses of tyrosine isomers on PK Day 1, and also associated with morning and evening doses of SM88, in patients with prostate cancer will be assayed.
Multi-dose steady state PK of all 4 components of SM88 in patients with prostate cancer. | Six months
  After approximately 2 weeks of daily dosing of SM88, the plasma concentrations of tyrosine isomers as well as the other 3 drugs of SM88 in patients with prostate cancer will be assayed.
Safety and tolerability of SM88 in patients with prostate cancer. | Six months
  Changes from baseline in blood work results and incidence of adverse events associated with treatment of SM88 in patients with prostate cancer.
Anti-cancer activities of SM88 in patients with prostate cancer. | Six Months
  Changes from baseline in CTCs, and PSA level per Prostate Cancer Working Group 3 (PCWG3) criteria and radiography per RECIST 1.1 criterial, stratified by circulating tumor cells (CTC) and other blood-based markers including lactate dehydrogenase (LDH), total alkaline phosphatase, bone-specific alkaline phosphatase, urine N-telopeptide, hemoglobin, and neutrophil:lymphocyte ratio (NLR).
Correlation of toxicity and efficacy with cutaneous hyperpigmentation | Six Months
  The incident and severity (as assessed by CTCAE v4.0) of treatment-related adverse events and anticancer activities of SM88 are correlated with the degree of cutaneous pigmentation (measured by quantitative image analysis of subject skin color). The total number of subjects with adverse events and efficacy with changes in skin pigmentation during treatment will be reported in aggregate. We will evaluate cutaneous pigmentation as a biomarker in the treatment of prostate cancer by SM88 and stratify pigmentation and known risk factors for outcome analysis.
Radiographic progression-free-survival (rPFS) | Six Months
  Duration of survival since treatment initiation with SM88 of study subjects who are without disease progression according to radiology, stratified by PSA level, CTC, and other blood-based markers (including LDH, total alkaline phosphatase, bone-specific alkaline phosphatase, urine N-telopeptide, hemoglobin, and NLR).
PSA doubling time before, during and after SM88 | Six Months
  PSA doubling time before, during and after SM88 treatment will be compared to evaluate disease progression rate associated with SM88 treatment.
Effect of SM88 on patient-reported outcomes including quality of life (as measured by the EORTC QLQ-30 and EORTC QLQ-PR25) in patients with prostate cancer. | Six Months
  Changes from baseline in the Quality-of-Life, as measured by EORTC QLQ-30 and QLQ-PR25, stratified by PSA level, CTC, and other blood-based markers (including LDH, total alkaline phosphatase, bone-specific alkaline phosphatase, urine N-telopeptide, hemoglobin, and NLR in patients with prostate cancer).
Effect of SM88 on performance status in patients with prostate cancer. | Six months
  Changes from baseline in the performance status (as measured by Eastern Cooperative Oncology Group (ECOG) score) in patients with prostate cancer.

OTHER OUTCOMES:
Cutaneous hyperpigmentation as a biomarker in the treatment of prostate cancer by SM88. | Six months
  Correlation between the anti-cancer activities of SM88 vs. the degree of cutaneous pigmentation (measured by quantitative image analysis of subject skin color). The total number of subjects with efficacy and changes in skin pigmentation during treatment will be reported in aggregate. We will evaluate cutaneous pigmentation as a biomarker for the efficacy of SM88 treatment in patients with prostate cancer.
Collection of lymphocyte counts as a biomarker for efficacy. | Six months
  The efficacy of SM88 will be correlated with lymphocyte counts. The total number of subjects with efficacy and lymphocyte counts during treatment will be reported in aggregate. We will evaluate lymphocyte counts as a biomarker for the efficacy of SM88 treatment in patients with prostate cancer.
Stratification of outcome with known risk factors for prostate cancer. | Six months
  Stratification of anticancer activities with known risk factors for prostate cancer.
Duration of time when a subsequent therapy is needed after treatment with SM88. | Six months
  The duration in time for another therapy due to recurrence of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Del Priore, MD, MPH, Study Director — Chief Medical Officer TYME Inc.
Locations (5):
- United States (5):
  - AdvanceMed Research, Lawrence, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - Montefiore Medical Center- Montefiore Medical Park, The Bronx, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steve Hoffman, et al. An open-label trial of SMK treatment of advanced metastatic cancer. J Clin Oncol 31, 2013 (suppl; abstr e22095)
- [Background] Steve Hoffman, et al. An Open-Label Trial of SMK Treatment of Advanced Metastatic Cancer. 18th World Congress on Controversies in Obstetrics, Gynecology & Infertility (COGI). 473-480, 2014 Monduzzi Editoriale | Proceedings.
- [Background] Avi Retter. Non-Hormonal Therapy for Recurrent Non-Metastatic Prostate Cancer. Oncology Times. 40(4):29-31, February 20, 2018.
- [Background] Del Priore G, Hoffman S. Timing of androgen-deprivation therapy in prostate cancer. Lancet Oncol. 2017 Nov;18(11):e633. doi: 10.1016/S1470-2045(17)30774-X. Epub 2017 Oct 31. No abstract available. PMID 29208387
- [Derived] Gartrell BA, Roach M 3rd, Retter A, Sokol GH, Del Priore G, Scher HI. Phase II trial of SM-88, a cancer metabolism based therapy, in non-metastatic biochemical recurrent prostate cancer. Invest New Drugs. 2021 Apr;39(2):499-508. doi: 10.1007/s10637-020-00993-4. Epub 2020 Sep 13. PMID 32924093